CLINICAL TRIAL: NCT01876264
Title: Crohn's Extent of Resection Trial (CERT): A Randomised Controlled Trial Comparing Anastomotic Disease Recurrence Following 2cm Versus 10cm Resection Margins for Patients With Ileocolic Crohn's Disease
Brief Title: Crohn's Extent of Resection Trial
Acronym: CERT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study abandoned
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CERT2013
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Crohn's Disease; Recurrence
Keywords: Colorectal surgery; Colonoscopy; Randomized controlled trial
MeSH Terms: conditions — Crohn Disease; Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extended resection (Experimental): Patients undergoing an extended resection are subjected to a traditional ileocolic resection with a 2cm macroscopically normal proximal margin. A further 8cm of ileum is then resected from the proximal margin prior to formation of the ileocolic anastomosis
  Interventions: Procedure: Extended resection
- Conventional resection (Active Comparator): Patients undergoing a traditional ileocolic resection for Crohn's disease with a 2cm proximal macroscopically disease-free margin
  Interventions: Procedure: Conventional resection

INTERVENTIONS:
Procedure: Extended resection
  Arms: Extended resection
Procedure: Conventional resection
  Arms: Conventional resection

SUMMARY:
The trial will investigate if removing an additional length of small bowel will result in lower risk of recurrence at the surgical join (anastomosis), thereby decreasing the need for further surgery in the future.

DETAILED DESCRIPTION:
The study will be conducted as a randomised controlled trial. The patient will be blinded to the procedure undertaken, as will the endoscopist performing the 6 month post operative colonoscopy. It is not possible to blind the operating team, for obvious reasons.

Patients undergoing elective or urgent ileocolic resection, both primary and redo resections, will be invited to participate in the trial. Randomisation will take place in the operating theatre after a conventional ileocolic resection has been performed. Those patients randomised to the modest resection (10cm margin) will have an additional 8cm of distal small bowel resected prior to the formation of the surgical anastomosis.

All patients will be seen in the colorectal clinic at approximately 6 weeks post operatively for their routine follow up appointment, as is current practice. A colonoscopy will be performed at 6 months post operatively to assess the anastomosis, in keeping with our current practice. Any additional follow up will be at the discretion of the colorectal or gastroenterological teams, in keeping with their clinical practice.

Patients recruited to the trial will not have any additional ongoing following up directly related to their trial participation. At 5 years following the recruitment of the a patient, the medical notes will be reviewed to identify those patients who have had symptomatic recurrence, further surgery and to assess the duration of medication-free interval following surgery.

Performing a colonoscopy at 6 months post operatively to assess the appearances of the surgical anastomosis will assess the primary endpoint. This will be performed by a senior gastroenterological trainee or consultant gastroenterologist who is familiar with assessment of post operative Crohn's disease and the Rutgeert's score. The appearances of the anastomosis will be scored, and biopsies taken from around the anastomosis to assess for microscopic changes. The use of the Rutgeert's score is widely accepted by the gastroenterological community as the standard assessment tool for post operative anastomotic disease recurrence in patients with Crohn's disease.

The duration of medication-free interval following resection will be assessed from review of the medical notes. This is clinically relevant to patients, as it has been previously shown that quality of life is improved in patients who do not have to take regular medication.

The duration of symptom-free interval will be assessed from review of the medical notes. This is clinically relevant to patients, as abdominal symptoms such as pain and bloating have a significantly deleterious effect on quality of life.

The duration of time to reoperation for Crohn's disease recurrence at the surgical anastomosis will be assessed from the clinical notes. This is of relevance to the patient population as well as the medical community. Crohn's disease commonly recurs, necessitating further surgery. Multiple operations resulting in resection of the bowel results in a reduction in the length of bowel available for absorption of nutrients from food. Ultimately, patients may develop short bowel syndrome. This requires total parenteral nutrition, with the associated risks this carries, and may require small bowel transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 16 years or above.
* Patients with ileocolic Crohn's disease requiring surgical resection

Exclusion Criteria:

* Patients unable to give informed consent
* Patients requiring formation of a stoma at the time of surgical resection
* Patients having less than 200cm of small bowel as assessed intra-operatively
* Simultaneous strictureplasty or small bowel resection
* Age <16 or >80

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06 (Estimated); Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Endoscopic recurrence | 6 months post operatively
  The primary objective of the study is to assess whether undertaking a modest ileocolic resection (10cm margins) leads to a reduction in the incidence of Crohn's disease recurrence at the surgical anastomosis as assessed by colonoscopy 6 months post operatively, when compared to a conventional ileocolic resection (2cm margin).

SECONDARY OUTCOMES:
Medication-free interval | 5 years post operatively
  To assess the impact of undertaking a modest ileocolic resection (10cm margin) on the duration of medication-free interval following surgery, with respect to disease-modifying drugs (e.g. azathioprine), when compared to a conventional ileocolic resection (2cm margin)
Symptom-free interval | 5 years post operatively
  To assess the impact of undertaking a modest ileocolic resection (10cm margin) on the duration of the symptom-free interval following surgery, when compared to a conventional ileocolic resection (2cm margin)
Time to reoperation | 5 years post operatively
  To assess the impact of undertaking a modest ileocolic resection (10cm margin) on the interval to reoperation (if clinically needed) for anastomotic recurrence when compared to a conventional ileocolic resection (2cm margin)
Extent of plexitis | 1 month postoperatively
  To assess the extent of plexitis through the length of macroscopically normal small bowel that is resected

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Lovegrove, MBBS MD FRCS, Principal Investigator — Worcestershire Acute Hospitals NHS Trust
Locations (1):
- Oxford University Hospitals NHS Trust, Oxford, United Kingdom